CLINICAL TRIAL: NCT03024307
Title: Evaluation of an Outpatient Pharmacy Clinical Services Program on Adherence and Clinical Outcomes Among Patients With Rheumatic Diseases
Brief Title: The Effect of OPCSP on Adherence and Clinical Outcomes Among Patients With Rheumatic Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Ting Li, Doctor, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OPCSP2016
Record Dates: First submitted 2016-10-11; First posted 2017-01-18 (Estimated); Last update posted 2021-03-04 (Actual); Status verified 2020-01

CONDITIONS: Rheumatic Diseases
Keywords: Pharmaceutical Care; Medication Adherence; Direct Costs
MeSH Terms: conditions — Rheumatic Diseases; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Involvement of pharmacists in improving medication (Experimental): Pharmacists involved care group. Tools used to improve medication adherence, (1)Patient medication guide (2)tailored Short Messaging Service (SMS) (3)Pharmaceutical follow-up
  Interventions: Other: pharmacists involved OPCSP
- usual care only (No Intervention): Patients were provided with usual care.

INTERVENTIONS:
Other: pharmacists involved OPCSP — This was an open labelled randomised study. Rheumatic diseases patients were recruited and arbitrarily divided into the intervention group (usual care plus OPCSP) and the non-intervention group (usual care only). Those enrolled in the research were scheduled for follow-up for eight consecutive visits. Improvements in lab results and direct costs were compared longitudinally (pre and post analysis) between the groups.
  Arms: Involvement of pharmacists in improving medication

SUMMARY:
This is a randomised trial on the efficacy of an Outpatient Pharmacy Clinical Services Program (OPCSP) on adherence and clinical outcomes among patients with rheumatic diseases.The purpose of this study is to evaluate:

1. rates of medication adherence in the OPCSP program compared with usual care in an integrated health care system.
2. total direct costs and clinical outcomes in the OPCSP program compared with usual care in an integrated health care system.

DETAILED DESCRIPTION:
This is a randomised trial on the efficacy of an Outpatient Pharmacy Clinical Services Program (OPCSP) on adherence and clinical outcomes among patients with rheumatic diseases.Three types of rheumatic diseases were included in the study, Systemic lupus erythematosus (SLE), Ankylosing spondylitis (AS), and Rheumatoid Arthritis(RA). The purpose of this study is to evaluate:

1. rates of medication adherence in the OPCSP program compared with usual care in an integrated health care system.
2. total direct costs and clinical outcomes in the OPCSP program compared with usual care in an integrated health care system.

ELIGIBILITY:
Inclusion Criteria:

* Willingness of the subject to participate in the study, proven by signing the informed consent;
* Systemic lupus erythematosus (SLE), as defined by meeting at least 4 of 11 classification criteria of American College of Rheumatology for the classification of systemic lupus erythematosus, either sequentially or coincidentally. The 4 criteria doesn't need to be present at the time of study enrollment;
* Patients fulfilled the American College of Rheumatology criteria for RA and AS;

Exclusion Criteria:

* Patients who are unwilling to sign the inform consent;
* Pregnancy or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Medication adherence in the OPCSP program compared with usual care | 12 months
  Medication adherence would be evaluated by the questionnaire survey, CQR19. Scores of medication adherence would be calculated.

SECONDARY OUTCOMES:
Changes in medical outcomes from baseline at each visit by EQ5D-3L | 12 months
  The influence of OPCSP on improving medical outcomes would be evaluated by EQ5D-3L. The TTO value would be compared between two arms
changes in direct costs from baseline at each visit | 12 months
  the influence of OPCSP on reducing direct costs

CONTACTS AND LOCATIONS:
Overall Officials: Shuang Ye, MD, Study Chair — RenJi Hospital
Locations (1):
- South Campus, Ren Ji Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang L, Luan W, Geng S, Ye S, Wang X, Qian L, Ding Y, Li T, Jiang A. Lack of patient education is risk factor of disease flare in patients with systemic lupus erythematosus in China. BMC Health Serv Res. 2019 Jun 13;19(1):378. doi: 10.1186/s12913-019-4206-y. PMID 31196083